CLINICAL TRIAL: NCT03268863
Title: Using the Cold Pressor Test to Assess Effectiveness of Low-Cost, Immersive Virtual Reality Therapy
Brief Title: Evaluating VR Therapy Using Cold Pressor Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janet Vittone (Other)
Responsible Party: Sponsor-Investigator, Janet Vittone, Consultant, General Internal Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-004181
Record Dates: First submitted 2017-07-28; First posted 2017-08-31 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: pain tolerance; perioperative pain; virtual reality therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Google Cardboard Virtual Reality headset running an interactive game
  Interventions: Device: Virtual Reality; Other: Cold Pressor
- Control (Sham Comparator): Powered down Google Cardboard Virtual Reality headset
  Interventions: Other: Cold Pressor

INTERVENTIONS:
Device: Virtual Reality — Google Cardboard virtual reality headset
  Arms: Virtual Reality
Other: Cold Pressor — A cold ice water bath for use in pain/discomfort simulation
  Other Names: Cold Pressor Test

SUMMARY:
This study is testing whether or not low-cost, virtual reality (VR) headsets for mobile phones can be used as a potential distractor from pain and thus would have clinical applications as a low-cost, non-pharmaceutical method to increase pain tolerance in patients undergoing painful or uncomfortable procedures. To do this, the investigators are asking volunteers to submerge their hand up to the wrist in cold water (Cold Pressor Test), either while playing an interactive virtual reality game on the headset, or while wearing a VR headset that is turned off as a control. The investigators will record the participants' tolerance to cold water as measured by how long the participants are able to keep their hand in the cold water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult Mayo Clinic students and employees

Exclusion Criteria:

* Participants who are known to be sensitive to VR technology and/or have undesirable reactions to VR technology (i.e. dizziness, motion sickness)
* Participants with significant alcohol/smoking histories, sickle cell anemia, history of previous myocardial infarction and/or coronary artery disease, malignant hypertension, metabolic
* dysfunctions, pregnancy, Raynaud's disease, epilepsy, severe mental disorders, chronic pain conditions, or diseases producing neuropathic pain
* Participants that have used drugs/alcohol the day prior to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Pain Tolerance | 10 minutes
  Likert Scale, 0-10

SECONDARY OUTCOMES:
Pain threshold | 10 minutes
  Onset of pain/discomfort as expressed verbally, in seconds and minutes
maximal pain | 10 minutes
  Likert scale
Nausea | 10 minutes
  modified Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Janet Vittone, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials